CLINICAL TRIAL: NCT00379873
Title: Chiropractic Adjustment on Physiological Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RD0606060021
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Healthy

INTERVENTIONS:
Device: ProAdjuster

SUMMARY:
This research is designed to study the effects of chiropractic adjustment on the physiological responses (EEG, EMG, HRV, skin temperature, and respiration) of college student and faculty population.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic subjects (without somatosensory peripheral pain) will be recruited in the study.

Exclusion Criteria:

Subjects with heart failure and any nervous system diseases will be excluded from the study. Additional exclusions include osteoporosis, pregnancy, diabetes, vascular insufficiency, and history of joint replacement therapy. Subjects under medical treatment, surgery and trauma within six months will be excluded

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
to understand the physiological response of a chiropractic adjustment

CONTACTS AND LOCATIONS:
Overall Officials: John Zhang, MD, PhD, Principal Investigator — Logan College of Chiropractic; Rodger Tepe, PhD, Study Director — Logan College of Chirppractic

REFERENCES:
- [Background] DeVocht JW, Pickar JG, Wilder DG. Spinal manipulation alters electromyographic activity of paraspinal muscles: a descriptive study. J Manipulative Physiol Ther. 2005 Sep;28(7):465-71. doi: 10.1016/j.jmpt.2005.07.002. PMID 16182019